CLINICAL TRIAL: NCT00974584
Title: A Phase Ib, Open-Label, Dose-Escalation Study of the Safety and Pharmacology Of PI3-Kinase Inhibitor GDC-0941 In Combination With Either Paclitaxel And Carboplatin (With or Without Bevacizumab) or Pemetrexed, Cisplatin, And Bevacizumab in Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: A Study of the Safety and Pharmacology Of PI3-Kinase Inhibitor GDC-0941 In Combination With Either Paclitaxel And Carboplatin (With or Without Bevacizumab) or Pemetrexed, Cisplatin, And Bevacizumab in Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GDC4628g; GO01303 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2009-09-08; First posted 2009-09-10 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
Keywords: NSCLC; PI3K; Avastin
MeSH Terms: interventions — 2-(1H-indazol-4-yl)-6-(4-methanesulfonylpiperazin-1-ylmethyl)-4-morpholin-4-ylthieno(3,2-d)pyrimidine; Bevacizumab; Carboplatin; Cisplatin; Paclitaxel; Pemetrexed

ARMS (4):
- GDC-0941+Paclitaxel+Carboplatin (Experimental): Bevacizumab-ineligible non-small cell lung cancer (NSCLC) participants may receive up to 6 cycles (21-day cycle) of combination chemotherapy with paclitaxel and carboplatin along with GDC-0941
  Interventions: Drug: GDC-0941; Drug: carboplatin; Drug: paclitaxel
- GDC-0941+Paclitaxel+Carboplatin+Bevacizumab (Experimental): Bevacizumab-eligible NSCLC particpants may receive up to 6 cycles of combination chemotherapy with paclitaxel and carboplatin along with GDC-0941 and bevacizumab.
  Interventions: Drug: GDC-0941; Drug: bevacizumab; Drug: carboplatin; Drug: paclitaxel
- GDC-0941+Pemetrexed+Cisplatin (Experimental): Bevacizumab-ineligible NSCLC participants may receive up to 6 cycles of combination chemotherapy with pemetrexed and cisplatin along with GDC-0941.\n
  Interventions: Drug: GDC-0941; Drug: bevacizumab; Drug: cisplatin; Drug: pemetrexed
- GDC-0941+Pemetrexed+Cisplatin+Bevacizumab (Experimental): Bevacizumab-eligible NSCLC participants may receive up to 6 cycles of combination chemotherapy with pemetrexed and cisplatin along with GDC-0941 and bevacizumab.\n
  Interventions: Drug: GDC-0941; Drug: bevacizumab; Drug: cisplatin; Drug: pemetrexed

INTERVENTIONS:
Drug: GDC-0941 — The GDC-0941 at a starting dose of 60 milligrams (mg) will be administered once daily orally for 14 consecutive days (Days 1 to 14) in 3-week cycles except for the first cycle that has Day 1 of single-agent GDC-0941 preceding Day 2 with combination chemotherapy.\n\n\n\n\n\n
Drug: bevacizumab — Bevacizumab 15 milligrams per kilograms (mg/kg) intravenously (IV) on Day 1 of every 3-week cycle.
  Arms: GDC-0941+Paclitaxel+Carboplatin+Bevacizumab; GDC-0941+Pemetrexed+Cisplatin; GDC-0941+Pemetrexed+Cisplatin+Bevacizumab
Drug: carboplatin — Carboplation IV on Day 1 of every 3-week cycle, at a dose to achieve an area under concentration time curve of 6 milligrams per milliliter*minute (mg/mL*min).\n
  Arms: GDC-0941+Paclitaxel+Carboplatin; GDC-0941+Paclitaxel+Carboplatin+Bevacizumab
Drug: cisplatin — Cisplatin 75 milligrams per square meter (mg/m^2) IV on Day 1 of every 3-week cycle.\n
  Arms: GDC-0941+Pemetrexed+Cisplatin; GDC-0941+Pemetrexed+Cisplatin+Bevacizumab
Drug: paclitaxel — Paclitaxel 200 mg/m^2 IV on Day 1 of every 3-week cycle.\n\n
  Arms: GDC-0941+Paclitaxel+Carboplatin; GDC-0941+Paclitaxel+Carboplatin+Bevacizumab
Drug: pemetrexed — Pemetrexed 500 mg/m^2 IV on Day 1 of every 3-week cycle.
  Arms: GDC-0941+Pemetrexed+Cisplatin; GDC-0941+Pemetrexed+Cisplatin+Bevacizumab

SUMMARY:
This is an open-label, multicenter, Phase Ib dose-escalation study to assess the safety, tolerability, and pharmacokinetics of oral (PO) GDC-0941 administered with one of three planned regimens: Arm A: paclitaxel and carboplatin in bevacizumab-ineligible NSCLC patients, Arm B: paclitaxel, carboplatin, and bevacizumab in bevacizumab-eligible NSCLC patients and Arm C: pemetrexed, cisplatin, and bevacizumab in bevacizumab-eligible, non-squamous NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented NSCLC with advanced disease (Stage IIIb not eligible for chemoradiotherapy or Stage IV or recurrent disease)
* Adequate organ function as assessed by laboratory tests
* Evaluable disease or disease measurable per Response Evaluation Criteria in Solid Tumors (RECIST)

Exclusion Criteria:

* More than one anti-cancer regimen (chemotherapy or radiotherapy) for advanced NSCLC prior to initiation of study treatment
* Any adjuvant or neoadjuvant anti-cancer therapy within a specified timeframe prior to first study treatment
* History of Grade >= 3 fasting hyperglycemia or diabetes requiring regular medication
* Active autoimmune disease, active infection requiring IV antibiotics, or other current uncontrolled illness
* History of clinically significant cardiac or pulmonary dysfunction
* History of malabsorption syndrome or other condition that would interfere with enteral absorption
* Clinically significant history of liver disease
* Any condition requiring full-dose anticoagulants, such as warfarin, heparin, or thrombolytic agents
* Known brain metastases that are untreated, symptomatic, or require therapy
* Pregnancy, lactation, or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2009-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicities (DLTs) | Days 1 to 22 of Cycle 1
Percentage of Participants with Adverse Events (AEs) | Up to approximately 5.5 years

SECONDARY OUTCOMES:
Maximum Plasma Concentration of Paclitaxel | Cycle 1 Day 2: Pre-paclitaxel infusion, end of paclitaxel infusion, 0.5, 1 and 2 hours post-paclitaxel infusion; Cycle 1 Day 3: Pre-GDC-0941 dose, 24 hours post-paclitaxel Day 2 infusion
Maximum Plasma Concentration of Carboplatin | Cycle 1 Day 2: Pre-carboplatin infusion, end of Carboplatin infusion, 0.5, 1.5 hours post-carboplatin infusion\n\n
Maximum Plasma Concentration of Pemetrexed | Cycle 1 Day 2: Pre-pemetrexed infusion, end of pemetrexed infusion, 1, 3 hours post-pemetrexed infusion; Cycle 1 Day 3: Pre-GDC-0941 dose, 24 hours post-pemetrexed Day 2 infusion\n\nd be "Yes".
Maximum Plasma Concentration of Cisplatin | Cycle 1 Day 2: Pre-cisplatin infusion, end of cisplatin infusion, 3 hours post-cisplatin infusion; Cycle 1 Day 3: Pre-GDC-0941 dose, 24 hours post-pemetrexed Day 2 infusion\n\n
Percentage of Participants with Objective Response (Complete or Partial Response), as Assessed Using Response Evaluation Criteria in Solid Tumors (RECIST) | Screening, Days 15 to 21 of Cycles 2, 4, 6, 9, and every 3 cycles thereafter (up to approximately 5.5 years)\n\n
Duration of Response, as Assessed Using RECIST\n\n\n | Screening, Days 15 to 21 of Cycles 2, 4, 6, 9, and every 3 cycles thereafter (up to approximately 5.5 years)
Progression-free Survival (PFS), as Assessed Using RECIST\n | Screening, Days 15 to 21 of Cycles 2, 4, 6, 9, and every 3 cycles thereafter (up to approximately 5.5 years)\n\n
Maximum Plasma Concentration of GDC-0941 | Cycle 1 Days 1 and 2: Pre-GDC-0941 dose, 1, 2, 3 and 4 hours post-GDC-0941 dose; Cycle 1 Days 3 and 9: Pre-GDC-0941 dose; 30 days after last dose of study treatment (up to approximately 5.5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (3):
- Buffalo, New York, United States
- Villejuif, France
- Groningen, Netherlands